CLINICAL TRIAL: NCT02573623
Title: Evaluation, of Innovative Tuberculosis Diagnostic Tests - Promoting Infant Health and Nutrition in Sub-Saharian Africa (PROMISE Consortium)
Brief Title: Evaluation of an Innovative Tuberculosis Diagnostic Test
Acronym: PROMISE-TB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS12293 PROMISE-TB
Record Dates: First submitted 2015-09-22; First posted 2015-10-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Tuberculosis; HIV
Keywords: Immunology diagnosis test; Children; Zambia
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine Serum Cell culture supernatant
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- HIV-infected children with confirmed TB: Hospitalized children with TB confirmed by culture or GeneXpert
- HIV-uninfected children aged<5 years with confirmed TB: Hospitalized children aged<5 years with TB confirmed by culture or GeneXpert
- HIV-uninfected children aged>4 years with confirmed TB: Hospitalized children aged>4 years with TB confirmed by culture or GeneXpert
- HIV-infected control children: Children hospitalized in the surgery ward without any evidence of tuberculosis infection
- HIV-uninfected controls aged <5 years: Children <5 years hospitalized in the surgery ward without any evidence of tuberculosis infection
- HIV-uninfected controls aged >4 years: Children >4 years hospitalized in the surgery ward without any evidence of tuberculosis infection

SUMMARY:
Diagnosis of tuberculosis (TB)in young children is a challenge due to atypical non-specific symptoms, difficulty to expectorate mucus, paucibacillary nature of pulmonary TB and low sensitivity of available diagnostic tools.

This project aims at evaluating two innovative immunological methods for diagnosing of active TB among HIV-infected and uninfected children.

DETAILED DESCRIPTION:
The study is designed as a prospective study for the evaluation of diagnostic tests.

Children admitted with probable TB based on clinical and radiological symptoms are recruited. Gastric lavage or sputum on two to three consecutive days will be collected as per routine practise. Active TB will be defined as a positive GeneXpert diagnostic test or MTB culture.

In addition, children with no sign of TB will be recruited to estimate the specificity of the diagnostic tests. These children will be recruited from the surgical ward of the hospital, and matched for age group and HIV status.

In all children, blood samples will be drawn and stored to perform quantiferon (R) and the new tests under evaluation.

The analysis will evaluate the sensitivity and specificity of the tests against the current gold standard (detection of Mycobacterium tuberculosis (MTB) in any specimen obtained from the patient). Identification of diagnosis algorithms, including these tests if they prove to be informative, will be elaborated and evaluated.

ELIGIBILITY:
Inclusion Criteria for tuberculosis cases:

* one of 4 clinical signs

  * persistent and unexplained cough
  * unexplained weight loss or failure to thrive
  * persistent and unexplained fever
  * persistent and unexplained lethargy or reduced playfulness
* chest X-Ray consistent with a tuberculosis infection
* an adenitis compatible with non-pulmonary tuberculosis Among these children only those with confirmed TB will be analysed for the primary outcome

Inclusion Criteria for controls:

* children without any of the signs and symptoms quoted above

Max Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 0 to 15 years with a definite diagnosis of tuberculosis infection, HIV-infected or uninfected.
  They will be matched on age and HIV status, to an equivalent number of children without any evidence of tuberculosis infection.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of children with tuberculosis who are correctly identified by a immunoenzymatic test for tuberculosis as having the condition | baseline
Proportion of tuberculosis negative children who are correctly identified as such by a immunoenzymatic test for tuberculosis | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Tuaillon, MD, PhD, Study Director — Université de Montpellier, France; Chipepo Kankasa, MD, PhD, Study Director — University of Zambia, Zambia; Philippe Van de Perre, MD, PhD, Study Chair — Université de Montpellier, France; Nicolas Nagot, MD, PhD, Principal Investigator — Université de Montpellier, France
Locations (1):
- Department of Paediatrics and Child Health, University Teaching Hospital.UNZA-SOM, Lusaka, Zambia